CLINICAL TRIAL: NCT04518722
Title: CT-Based Changes in Bone and Marrow Among Patients on Oral Steroids
Status: Recruiting | Type: Observational
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Punam K Saha, Professor, University of Iowa
Other Study IDs: 202009045
Record Dates: First submitted 2020-08-14; First posted 2020-08-19 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Asthma; Bone Density, Low; Oral Steroid-Dependent Asthma (Disorder)
Keywords: Glucocorticoid; Corticosteroid
MeSH Terms: conditions — Asthma; Bone Diseases, Metabolic | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Radiation: CT Scan — Dual-energy mid-tibia CT, high-resolution single energy MDCT imaging of the distal tibia (ankle), and low radiation hip CT scans
  Other Names: CAT Scan
Radiation: DXA Scan — Basic DXA scans will be performed to measure areal BMD and body composition measures at the whole body, spine, and hip
  Other Names: Bone Density Scan
Other: Steroid Intake Questionnaire — Questionnaire designed to quantify lifetime oral glucocorticoid intake

SUMMARY:
The goal of this study is to assess the feasibility of emerging CT-based tools to measure changes in central and peripheral bone density, micro-structure, and marrow adipose tissue (MAT) among patients treated with oral steroids.

DETAILED DESCRIPTION:
This study aims to prove that emerging CT-based tools are suitable to measure changes in central and peripheral bone density, geometry, micro-structure, and marrow adipose tissue (MAT) among patients treated with oral steroids. To do this, investigators will recruit 10 non-smokers (defined as < 10 pack-year smoking history) age 25-45 years with a diagnosis of severe, persistent asthma who either chronically use oral steroids or do not use any oral steroids. Participants will undergo dual-energy X-ray absorptiometry (DXA), dual-energy mid-tibia CT, high-resolution single-energy ankle CT, and low-radiation hip CT scans at baseline and 6-month follow-up visits. The images obtained will be used to analyze cross-sectional differences in central and peripheral bone density, geometry, micro-structure, and MAT between patients using oral steroids versus those who do not use any oral steroids. Differences in imaging at baseline and six-month follow visits will be used to analyze longitudinal bone changes among patients with oral steroid treatment.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion (all subjects):

  * Diagnosis of severe, persistent asthma (defined as using both a long-acting beta-agonist AND a high-dose inhaled steroid)
  * Age 25-45
* Inclusion (oral steroid group):

  * Chronic treatment with oral steroids for at least 45 days but less than 1 year

Exclusion Criteria:

* Exclusion (all subjects):

  * Pregnant or breastfeeding
  * History of any cancer, excluding non-melanoma skin cancer
  * Currently receiving dialysis
  * History of any lower extremity fracture
  * Hip or knee replacement
  * Non-ambulatory
  * Greater than 10 pack-year smoking history
  * BMI > 50
  * Age < 25 or > 45
  * Current or past use of FDA-approved medication for osteoporosis:

Bisphosphonates (Alendronate/Fosamax, Ibandronate/Boniva, Risedronate/Actonel/Atelvia, Zoledronic Acid/Reclast) Calcitonin (Fortical, Miacalcin) Selective Estrogen Receptor Modulator (Raloxifene/Evista) Parathyroid Hormone Analogue (Teriparatide/Forteo) Monoclonal Antibody (Denosumab/Prolia)

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: We plan to enroll 12 subjects, divided into two groups of 6. We will recruit 6 subjects with a diagnosis of severe, persistent asthma who have been taking oral GCs for 1.5-11 months. We will also recruit 6 subjects with a diagnosis of severe, persistent asthma who have not used any oral GCs in the last 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Marrow Adipose Tissue | Baseline
  Marrow adipose tissue fraction at 14-16% location of the distal tibia from DECT ankle scans will be computed and compared between oral steroid and control groups.
Cortical Bone Density | Baseline
  Cortical bone density will be computed through CT scanning at 4-6% and 12-14% distal tibia locations and compared between oral steroid and control groups.
Peripheral Bone Density | Baseline
  Peripheral bone density will be computed through CT scanning at 4-6% and 12-14% distal tibia locations and compared between oral steroid and control groups.
Bone Geometry and Microstructure | Baseline
  Hip MDCT scans will be used compute volumetric bone mineral density (vBMD) measures over trabecular and cortical bone compartments at femoral head, femoral neck, greater trochanter, and lesser trochanter. These measurements will be compared between oral steroid and control groups.
DXA Body Composition Analysis (fat mass, lean mass, percent fat) | Baseline
  DXA scans will be used to acquire bone and soft tissue measures that will allow for the calculation of body composition measures, which will then be compared between oral steroid and control groups.
DXA Bone Mineral Density | Baseline
  DXA Bone Mineral Density score will be obtained using standard DXA scans and compared between oral steroid and control groups.

SECONDARY OUTCOMES:
Marrow Adipose Tissue | Change from baseline to 6-month follow up visit
  Marrow adipose tissue fraction at 14-16% location of the distal tibia from DECT ankle scans will be computed and evaluated over time in the oral steroid group.
Cortical Bone Density | Change from baseline to 6-month follow up visit
  Cortical bone density will be computed through CT scanning at 4-6% and 12-14% distal tibia locations and evaluated over time in the oral steroid group.
Peripheral Bone Density | Change from baseline to 6-month follow up visit
  Peripheral bone density will be computed through CT scanning at 4-6% and 12-14% distal tibia locations and evaluated over time in the oral steroid group.
Bone Geometry and Microstructure | Change from baseline to 6-month follow up visit
  Hip MDCT scans will be used compute volumetric bone mineral density (vBMD) measures over trabecular and cortical bone compartments at femoral head, femoral neck, greater trochanter, and lesser trochanter. Changes in these measurements from baseline to 6-month follow up visits will be computed for the oral steroid group.
DXA Body Composition Analysis (fat mass, lean mass, percent fat) | Change from baseline to 6-month follow up visit
  DXA scans will be used to acquire bone and soft tissue measures that will allow for the calculation of body composition measures. Change over time from baseline to 6-month follow up visit will be computed for the oral steroid group.
DXA Bone Mineral Density | Change from baseline to 6-month follow-up visit
  DXA Bone Mineral Density score will be obtained using standard DXA scans. These scores will be compared at baseline and 6-month follow up visits for the oral steroid group.

CONTACTS AND LOCATIONS:
Overall Officials: Punam K Saha, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Staa TP, Leufkens HG, Abenhaim L, Zhang B, Cooper C. Use of oral corticosteroids and risk of fractures. J Bone Miner Res. 2000 Jun;15(6):993-1000. doi: 10.1359/jbmr.2000.15.6.993. PMID 10841167
- [Background] Canalis E, Mazziotti G, Giustina A, Bilezikian JP. Glucocorticoid-induced osteoporosis: pathophysiology and therapy. Osteoporos Int. 2007 Oct;18(10):1319-28. doi: 10.1007/s00198-007-0394-0. Epub 2007 Jun 14. PMID 17566815
- [Background] Clowes JA, Peel N, Eastell R. Glucocorticoid-induced osteoporosis. Curr Opin Rheumatol. 2001 Jul;13(4):326-32. doi: 10.1097/00002281-200107000-00015. PMID 11555737
- [Background] Wehrli FW, Saha PK, Gomberg BR, Song HK, Snyder PJ, Benito M, Wright A, Weening R. Role of magnetic resonance for assessing structure and function of trabecular bone. Top Magn Reson Imaging. 2002 Oct;13(5):335-55. doi: 10.1097/00002142-200210000-00005. PMID 12464746
- [Background] Barger-Lux MJ, Recker RR. Bone microstructure in osteoporosis: transilial biopsy and histomorphometry. Top Magn Reson Imaging. 2002 Oct;13(5):297-305. doi: 10.1097/00002142-200210000-00002. PMID 12464743
- [Background] Bell KL, Loveridge N, Power J, Garrahan N, Meggitt BF, Reeve J. Regional differences in cortical porosity in the fractured femoral neck. Bone. 1999 Jan;24(1):57-64. doi: 10.1016/s8756-3282(98)00143-4. PMID 9916785
- [Background] Kleerekoper M, Villanueva AR, Stanciu J, Rao DS, Parfitt AM. The role of three-dimensional trabecular microstructure in the pathogenesis of vertebral compression fractures. Calcif Tissue Int. 1985 Dec;37(6):594-7. doi: 10.1007/BF02554913. PMID 3937580
- [Background] Legrand E, Chappard D, Pascaretti C, Duquenne M, Krebs S, Rohmer V, Basle MF, Audran M. Trabecular bone microarchitecture, bone mineral density, and vertebral fractures in male osteoporosis. J Bone Miner Res. 2000 Jan;15(1):13-9. doi: 10.1359/jbmr.2000.15.1.13. PMID 10646109
- [Background] Legrand E, Audran M, Guggenbuhl P, Levasseur R, Chales G, Basle MF, Chappard D. Trabecular bone microarchitecture is related to the number of risk factors and etiology in osteoporotic men. Microsc Res Tech. 2007 Nov;70(11):952-9. doi: 10.1002/jemt.20501. PMID 17661392
- [Background] Moore RJ, Durbridge TC, McNeil PJ, Parkinson IH, Need AG, Vernon-Roberts B. Trabecular spacing in post-menopausal Australian women with and without vertebral fractures. Aust N Z J Med. 1992 Jun;22(3):269-73. doi: 10.1111/j.1445-5994.1992.tb02124.x. PMID 1386728
- [Background] Mosekilde L. Consequences of the remodelling process for vertebral trabecular bone structure: a scanning electron microscopy study (uncoupling of unloaded structures). Bone Miner. 1990 Jul;10(1):13-35. doi: 10.1016/0169-6009(90)90046-i. PMID 2397325
- [Background] Parfitt AM, Mathews CH, Villanueva AR, Kleerekoper M, Frame B, Rao DS. Relationships between surface, volume, and thickness of iliac trabecular bone in aging and in osteoporosis. Implications for the microanatomic and cellular mechanisms of bone loss. J Clin Invest. 1983 Oct;72(4):1396-409. doi: 10.1172/JCI111096. PMID 6630513
- [Background] Parfitt AM. Implications of architecture for the pathogenesis and prevention of vertebral fracture. Bone. 1992;13 Suppl 2:S41-7. doi: 10.1016/8756-3282(92)90196-4. PMID 1627414
- [Background] Recker RR. Architecture and vertebral fracture. Calcif Tissue Int. 1993;53 Suppl 1:S139-42. doi: 10.1007/BF01673423. PMID 8275368
- [Background] Vesterby A, Gundersen HJ, Melsen F, Mosekilde L. Marrow space star volume in the iliac crest decreases in osteoporotic patients after continuous treatment with fluoride, calcium, and vitamin D2 for five years. Bone. 1991;12(1):33-7. doi: 10.1016/8756-3282(91)90052-k. PMID 2054234
- [Background] Stone KL, Seeley DG, Lui LY, Cauley JA, Ensrud K, Browner WS, Nevitt MC, Cummings SR; Osteoporotic Fractures Research Group. BMD at multiple sites and risk of fracture of multiple types: long-term results from the Study of Osteoporotic Fractures. J Bone Miner Res. 2003 Nov;18(11):1947-54. doi: 10.1359/jbmr.2003.18.11.1947. PMID 14606506
- [Background] Li C, Jin D, Chen C, Letuchy EM, Janz KF, Burns TL, Torner JC, Levy SM, Saha PK. Automated cortical bone segmentation for multirow-detector CT imaging with validation and application to human studies. Med Phys. 2015 Aug;42(8):4553-65. doi: 10.1118/1.4923753. PMID 26233184
- [Background] Saha PK, Liu Y, Chen C, Jin D, Letuchy EM, Xu Z, Amelon RE, Burns TL, Torner JC, Levy SM, Calarge CA. Characterization of trabecular bone plate-rod microarchitecture using multirow detector CT and the tensor scale: Algorithms, validation, and applications to pilot human studies. Med Phys. 2015 Sep;42(9):5410-25. doi: 10.1118/1.4928481. PMID 26328990
- [Background] Chen C, Zhang X, Guo J, Jin D, Letuchy EM, Burns TL, Levy SM, Hoffman EA, Saha PK. Quantitative imaging of peripheral trabecular bone microarchitecture using MDCT. Med Phys. 2018 Jan;45(1):236-249. doi: 10.1002/mp.12632. Epub 2017 Nov 23. PMID 29064579
- [Background] Rosen CJ, Bouxsein ML. Mechanisms of disease: is osteoporosis the obesity of bone? Nat Clin Pract Rheumatol. 2006 Jan;2(1):35-43. doi: 10.1038/ncprheum0070. PMID 16932650
- [Background] Bredella MA, Gill CM, Gerweck AV, Landa MG, Kumar V, Daley SM, Torriani M, Miller KK. Ectopic and serum lipid levels are positively associated with bone marrow fat in obesity. Radiology. 2013 Nov;269(2):534-41. doi: 10.1148/radiol.13130375. Epub 2013 Jul 16. PMID 23861502
- [Background] Bredella MA, Daley SM, Kalra MK, Brown JK, Miller KK, Torriani M. Marrow Adipose Tissue Quantification of the Lumbar Spine by Using Dual-Energy CT and Single-Voxel (1)H MR Spectroscopy: A Feasibility Study. Radiology. 2015 Oct;277(1):230-5. doi: 10.1148/radiol.2015142876. Epub 2015 May 19. PMID 25988401